CLINICAL TRIAL: NCT04023630
Title: An Open-label, Randomized, Controlled, Multicenter Study to Evaluate DUAL Antithrombotic Therapy With Rivaroxaban Plus Ticagrelor vs. Rivaroxaban Plus Clopidogrel in Patients With Atrial Fibrillation and Acute Coronary Syndrome
Brief Title: DUAL Antithrombotic Therapy in Patients With AF and ACS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Jian'an Wang,MD,PhD, President of Second Affiliated Hospital, School of Medicine, Zhejiang University & Chief of Cardiology, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHZJU CT013
Record Dates: First submitted 2019-07-16; First posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Atrial Fibrillation; Acute Coronary Syndromes
MeSH Terms: conditions — Atrial Fibrillation; Acute Coronary Syndrome | interventions — Rivaroxaban; Tablets; Clopidogrel; Purinergic P2Y Receptor Antagonists; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rivaroxaban plus ticagrelor (Experimental): rivaroxaban 15 mg (or 10 mg for subjects with moderate renal impairment) once daily plus ticagrelor 90 mg tablet twice daily for 12 months
  Interventions: Drug: Rivaroxaban 15 MG Oral Tablet; Drug: Ticagrelor 90 MG Oral Tablet
- rivaroxaban plus clopidogrel (Active Comparator): rivaroxaban 15 mg (or 10 mg for subjects with moderate renal impairment) once daily plus clopidogrel 75 mg tablet once daily for 12 months
  Interventions: Drug: Rivaroxaban 15 MG Oral Tablet; Drug: Clopidogrel 75 Mg Oral Tablet

INTERVENTIONS:
Drug: Rivaroxaban 15 MG Oral Tablet — One 15 mg tablet once daily for up to twelve months
  Other Names: Xarelto
Drug: Clopidogrel 75 Mg Oral Tablet — One 75 mg tablet once daily for up to twelve months
  Other Names: P2Y12 antagonists
  Arms: rivaroxaban plus clopidogrel
Drug: Ticagrelor 90 MG Oral Tablet — One 90 mg tablet twice daily for up to twelve months
  Other Names: P2Y12 antagonists
  Arms: rivaroxaban plus ticagrelor

SUMMARY:
The study aims to show inferiority of rivaroxaban plus ticagrelor when compared to rivaroxaban plus clopidogrel in terms of safety. Safety will be determined by comparing the rates of death or ischemic event-including myocardial infarction, definite or probable stent thrombosis, stroke, or urgent revascularization.

DETAILED DESCRIPTION:
The main objective of this study is to compare a Dual Antithrombotic Therapy (DAT) regimen of rivaroxaban plus ticagrelor with rivaroxaban plus clopidogrel in Patients With Non Valvular Atrial Fibrillation (NVAF) and Acute Coronary Syndrome. The study aims to show inferiority of rivaroxaban plus ticagrelor when compared to rivaroxaban plus clopidogrel in terms of safety. Safety will be determined by comparing the rates of death or ischemic event-including myocardial infarction, definite or probable stent thrombosis, stroke, or urgent revascularization.

ELIGIBILITY:
Inclusion Criteria:

1. Adults with either active or a history of non-valvular atrial fibrillation or flutter with the planned or existing use of an oral anticoagulant for prophylaxis of thromboembolism. In addition, subjects must have had an acute coronary syndrome
2. Planned use of antiplatelet agents for at least 12 months
3. Males and Females ≥ 18 years of age
4. Women of childbearing potential must have a negative serum or urine pregnancy test within 24 hours prior to the start of study drug

Exclusion Criteria:

1. Conditions other than atrial fibrillation that require chronic anticoagulation. (e.g. prosthetic mechanical heart valve)
2. Severe renal insufficiency (serum creatinine > 2.5 mg/dL or a calculated creatinine clearance < 30 mL/min
3. Patients with a history of intracranial hemorrhage
4. Patients have had or will undergo Coronary arterial bypass graft (CABG) for their index acute coronary syndrome (ACS) event
5. Patients with known ongoing bleeding and patients with known coagulopathies
6. Any contraindications or allergies to rivaroxaban, or to intended P2Y12 antagonists
7. Have a history of stroke or Transient Ischemic Attack (TIA)
8. Have known significant liver disease or liver function test (LFT) abnormalities
9. Have any severe condition that would limit life expectancy to less than 12 months

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
The composite endpoints of death and ischemic events | one year
  The composite endpoints of death and ischemic events (stroke, myocardial infarction, stent thrombosis, urgent revascularization )

SECONDARY OUTCOMES:
Clinically significant bleeding | one year
  Clinically significant bleeding is a composite of Thrombolysis in Myocardial Infarction (TIMI) major bleeding, minor bleeding, and bleeding requiring medical attention (BRMA)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Jiang, PhD, Study Director — Second Affiliated Hospital Zhejiang University School of Medicine